CLINICAL TRIAL: NCT04699422
Title: Serratus Anterior Plane Block Versus Standard of Care After Totally Endoscopic Aortic Valve Replacement: a Double-blinded Randomized Controlled Trial.
Brief Title: Serratus Anterior Plane Block Versus Standard of Care After Totally Endoscopic Aortic Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principal Investigator, Jessa Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JessaH_SAPblock
Record Dates: First submitted 2020-11-30; First posted 2021-01-07 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Analgesia; Surgery; Cardiac Disease
MeSH Terms: conditions — Agnosia; Heart Diseases | interventions — Pirinitramide

STUDY DESIGN:
Intervention Model Description: This trial is designed as a mono-center, double-blinded, prospective, randomized controlled superiority trial comparing 2 groups of patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Patients in the experimental group will receive the serratus anterior plane block combined with postoperative PCIA with Piritramide.
  Interventions: Procedure: Serratus anterior plane block; Drug: PCIA with Piritramide
- Control group (Sham Comparator): Patients in the control group will receive postoperative PCIA with Piritramide.
  Interventions: Drug: PCIA with Piritramide

INTERVENTIONS:
Procedure: Serratus anterior plane block — The needle will be introduced in-plane from supero-anterior to postero-inferior until the needle tip is positioned in the plane underneath the serratus muscle (deep compartment). Under continuous ultrasound guidance,30 cc Bupivacaine 0.25% will be injected in the deep compartment. After the deep component of the SAP is completed, the needle will be withdrawn to the subcutaneous tissues. The needle will be flattened and advanced in-plane to the plane superficial to the serratus muscles. 10 cc Bupivacaine 0.25% will be injected superficial to the serratus muscles after correct placement of the needle tip is confirmed on ultrasound
  Arms: Experimental group
Drug: PCIA with Piritramide — A patient controlled intravenous analgesia system (IVAC PCAM®, Cardinal Health or CADD pump) with piritramide (Dipidolor®, Janssen) using following settings: bolus 2 mg and lockout interval 15 min.
  Other Names: PCIA with Dipidolor

SUMMARY:
The aim of this study is to assess and compare the efficacy of a serratus anterior plane (SAP) block and our current pain protocol (Patient Controlled Intravenous Analgesia with opioids) in the prevention and treatment of acute postoperative pain after totally endoscopic aortic valve replacement (AVR) surgery.

DETAILED DESCRIPTION:
During the last two decades, cardiac surgical techniques changed dramatically. Evidence for good short and long-term outcome after endovascular and minimally invasive procedures is rising. The goal of avoiding sternotomy is earlier patient recovery without compromising safety. Therefore, enhanced recovery after surgery (ERAS) protocols have been implemented to aim for early extubation and ambulation. Analgesic regimens after cardiac surgery did not change significant however. Opioids remain the cornerstone of analgesia in the postoperative cardiac surgical care units, despite known side effects as nausea, constipation and risk for addiction. Neuraxial anesthetic techniques after cardiac surgery have been studied and validated to reduce opioid consumption. Their implementation in clinical practice however remains limited for two reasons. First, heparinization is required for cardiac surgery, which increases the risk neuraxial hematoma after neuraxial anesthesia, leading to deleterious complications as paraplegia. Secondly, neuraxial anesthesia induces orthosympathicolysis, enhancing vasoplegia after cardiac surgery. However, fascial plane blocks in cardiac surgery since peripheral blocks do not induce sympathicolysis and consequences of chest wall hematoma are limited.

In 2013, Blanco described the serratus anterior plane (SAP) block as an analgesic option for chest wall surgery. In this fascial plane block, local anesthetics are injected in the plane beneath the anterior serratus muscle and in the plane between latissimus dorsi and serratus anterior in an ultrasound guided manner. SAP block provides analgesia in dermatomes T2-T9. Recently, successful analgesia after SAP block has been demonstrated for soft tissue chest wall surgery, thoracotomy and rib fractures. No major side effects were reported. More specifically, no sympatholytic effects or chest wall hematoma were observed. However, up to now no prospective studies assessing the analgesic efficacy of SAP block after cardiac surgery are published. Two retrospective studies show conflicting results. Berthoud et al. retrospectively compared SAP block to continuous wound infusion after different types of minimally invasive cardiac surgery (MICS) and found reduced morphine consumption as well as shorter intensive care and hospital length of stay after SAP block. In contrast, Moll et al. found no difference in opioid consumption between SAP block and no block in patients after robotic coronary artery bypass grafting (rCABG). The authors comment they only performed the deep component of the SAP block, and some surgical entry points were outside dermatomes T2-T7.

Totally endoscopic aortic valve replacement (AVR) is a novel minimally invasive cardiosurgical technique. Surgical incision is made anteriorly in intercostal space two on the right hemithorax. Since intercostal space two is innervated by dermatomes T2-T3, somatic analgesia can be obtained with SAP block. In addition with a favorable safety profile and a minimal/non-existent risk of evoking sympatholytic effects, a SAP block may be a suitable analgesic technique to prevent/minimize postoperative pain after totally endoscopic AVR surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective aortic valve replacement surgery via right anterolateral thoracotomy
* Adult patients (minimally 18 years old)
* EuroScore ii < 3%
* Bodyweight > 50 kg

Exclusion Criteria:

* Refusal to participate
* Inability to communicate due to language or neurologic barriers
* Inability to control and self-administer opioids with PCIA or to comprehend the NRS pain score due to confusion or learning difficulties
* Chronic use of opioids
* Chronic use of analgesic antidepressants and/or antiepileptics
* History of major trauma or surgery to right chest wall
* History of chronic pain at right chest wall
* Allergy to opioids and/or local anesthetics
* Allergy to acetaminophen
* Morbid obesity (BMI > 35)
* Pregnancy
* Peroperative events compromising early postoperative recovery (aortic dissection, systolic anterior motion of the mitral valve, cardiac tamponade, ..)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Cumulative opioid consumption by patient-controlled intravenous analgesia (PCIA) | 24 hours after performing the SAP block
  Piritramide consumption (mg) will be directly read from the PCIA-system after 24 hours.

SECONDARY OUTCOMES:
Opioid consumption during predetermined time intervals after surgery | Every 4 hours until 24 hours after placement of the SAP block
  Piritramide consumption (mg) will be directly read from the PCIA-system at predetermined time intervals after performing the SAP block.
Opioid free patients first 24 postoperative hours | First 24 hours
  Number of patients that do not require any opioids within the first 24 hours after surgery.
Opioid free patients during hospital length of stay | Through study completion, an average of 7 days
  Number of patients that do not require any opioids during the hospital length of stay
Postoperative pain score in rest | 4, 8, 12, and 24 hours after performing the SAP block and at postoperative day 7.
  The postoperative pain on the surgical site is evaluated based on an 11-points numeric scale (Numerical Rating Sale - NRS) where 0 = no pain and 10 = worst pain ever.
Quality of recovery after totally endoscopic aortic valve replacement | Postoperative days 2 and 7
  Quality of recovery will be assessed via the 5-Dimensional European Quality of Life (EQ5D) and 36-Item Short Form Health Survey (SF-36) questionnaires concerning mobility, self care, daily activities and pain.
Overall patient satisfaction with analgesic therapy | 24 hours after performing the serratus anterior plane block at postoperative day 1
  Overall patient satisfaction with analgesic therapy will be assessed with an 11-point Numeric Rating Scale (where 0 = not satisfied at all and 10 = extremely satisfied).
Postoperative nausea and vomiting (PONV) | 24 hours after performing the serratus anterior plane block at postoperative day 1
  The simplified postoperative nausea and vomiting (PONV) impact scale will be used to assess PONV. The scale ranges from 0 to 6, where 0 means no nausea/vomiting. Clinically important PONV will be defined as a score of 5 or more.
Constipation | Until postoperative day 7
  Time to first defecation (postoperative days) or need for laxatives during hospital stay.
Time to extubation | Throughout study completion, an average of 7 days
  Time from arrival to the ICU until extubation in minutes.
ICU length of stay | Until postoperative day 7
  Time from arrival to the ICU until meeting discharge criteria to the ward in postoperative hours.
Hospital length of stay | Through study completion, an average of 7 days
  Time to discharge out of the hospital in postoperative days (day of surgery = day 0)
Pneumonia | Until postoperative day 7
  Defined as empirical antibiotic therapy for suspicion of pneumonia during hospital stay, in number of patients.
Duration of vasopressor infusion | Until postoperative day 7
  Time from arrival to the ICU until full weaning from vasoactive substances (eg norepinephrine) in minutes. Patients not requiring any vasopressors will be excluded from this secondary outcome parameter.
Subcutaneous emphysema | 24 hours after performing the serratus anterior plane block at postoperative day 7
  Number of patients suffering subcutaneous emphysema. All patients will be investigated 24h after performing the SAP block (or control) by a blinded assessor.
Number of patients with new onset perioperative atrial fibrillation (POAF) | Until postoperative day 7
  Number of patients suffering witnessed (ECG recorded) POAF and patients with history of (paroxysmal) atrial fibrillation will not be taken into account for this secondary outcome parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Bjorn Stessel, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vandenbrande J, Jamaer B, Stessel B, van Hilst E, Callebaut I, Yilmaz A, Packle L, Sermeus L, Blanco R, Jalil H. Serratus plane block versus standard of care for pain control after totally endoscopic aortic valve replacement: a double-blind, randomized controlled, superiority trial. Reg Anesth Pain Med. 2024 Jun 3;49(6):429-435. doi: 10.1136/rapm-2023-104439. PMID 37597856